CLINICAL TRIAL: NCT00006399
Title: Estrogen Modulation Effects on Cholinergic Function in Normal Post-Menopausal Women and Patients With Alzheimer's Disease
Brief Title: Effects of Estrogen on Memory in Post-Menopausal Women and Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Alzheimer's Association (Other); Pfizer (Industry); Eisai Inc. (Industry)
Responsible Party: Paul A. Newhouse, M.D, Department of Psychiatry, University of Vermont College of Medicine
Organization: National Institute on Aging (NIA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: IA0023; 2R56AG021476 (NIH)
Record Dates: First submitted 2000-08-18; First posted 2000-08-21 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Estrogen therapy; Post-menopausal women
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; Estrogens; Progesterone

INTERVENTIONS:
Drug: Donepezil
Drug: Estrogen
Drug: Progesterone

SUMMARY:
The goal of this study is to examine whether the administration of estrogen to post-menopausal women and women with mild to moderate Alzheimer's disease will enhance their memory and their capacity for learning.

DETAILED DESCRIPTION:
Estrogen (EST) may have significant benefits in preserving cognitive functioning in normal aging after menopause and in decreasing the incidence of Alzheimer's disease (AD). On a molecular level, EST has effects on a variety of cholinergic neuronal and receptor-mediated mechanisms that may be responsible for these beneficial effects. These neurons have critical relevance for the development of age-related cognitive changes and dementing disorders. However, little is known about the clinical relevance of EST-cholinergic interactions, either in normal aging or in AD.

The primary goal of this study is to test the hypothesis that three months of administration of EST to 1) normal post-menopausal women, and 2) female patients with mild-moderate AD who are concurrently treated with anticholinesterase therapy (donepezil), will positively change or blunt the negative and behavioral effects of drugs that block central cholinergic receptors (both muscarinic and nicotinic). Participants will be blindly placed on EST or placebo for three months each. After each three month period, they will be cognitively assessed after receiving single doses of the cholinergic antagonists scopolamine and mecamylamine. These results will have direct implications for the use of EST in post-menopausal women as well as interactive treatment with cholinergic drugs for AD. Researchers plan to recruit a total of 45 women (30 healthy, and 15 patients with AD).

NOTE: This study is only recruiting participants with Alzheimer's Disease at this time.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers and women with mild Alzheimer's disease:
* Non-smoker
* No use of Hormone Replacement Therapy for at least one year
* No menses for at least one year
* Normal mammogram within the last year
* minimum age is 45 for patients with Alzheimer's disease; 50 for normal volunteers
* Maximum age is 85 for patients with Alzheimer's disease; there is no maximum age for normal volunteers.

Exclusion Criteria:

* Women who are currently taking estrogen therapy.
* Women who are smokers.
* Women who have had breast cancer.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 1999-09; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Newhouse, M.D., Principal Investigator — Memory Center, Department of Psychiatry, University of Vermont College of Medicine
Locations (1):
- Clinical Neuroscience Research Unit, University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Background] Newhouse PA, Potter A, Corwin J, Lenox R. Acute nicotinic blockade produces cognitive impairment in normal humans. Psychopharmacology (Berl). 1992;108(4):480-4. doi: 10.1007/BF02247425. PMID 1410163
- [Background] Newhouse PA, Potter A, Corwin J, Lenox R. Age-related effects of the nicotinic antagonist mecamylamine on cognition and behavior. Neuropsychopharmacology. 1994 Apr;10(2):93-107. doi: 10.1038/npp.1994.11. PMID 8024677
- [Background] Newhouse PA, Potter A, Corwin J, Lenox, R. Effects of nicotinic cholinergic agents on cognitive functioning in Alzheimer's and Parkinson's disease. Drug Development Research 38:278-289, 1996.
- See also: University of Vermont, Clinical Neuroscience Research Unit — http://www.uvm.edu/~cnru/